CLINICAL TRIAL: NCT07263035
Title: Urine Sodium-Driven Diuretic Adjustment Strategy in Acute Decompensated Heart Failure
Acronym: US-DASH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lakeland Regional Health Systems, Inc. (Other)
Responsible Party: Principal Investigator, Anas Bizanti, MD, Associate Program Director, Internal Medicine Residency - Principal Investigator, Lakeland Regional Health Systems, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025_001
Record Dates: First submitted 2025-11-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Heart Failure - NYHA II - IV; Heart Failure Acute; Acute Heart Failure (AHF)
Keywords: Urine sodium; Diuretics; Lasix; heart failure; Acute CHF; acute HFrEF; Acute HFpEF; Natriuresis
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): Traditional diuretic dosing adjustment per provider
  Interventions: Drug: Furosemide intravenous solution
- 50 mmol/L urine sodium (Experimental): Diuretics will be titrated to achieve a urine sodium concentration of 50 mmol/L
  Interventions: Drug: Furosemide intravenous solution
- 85 mmol/L urine sodium (Experimental): Diuretics will be titrated to achieve a urine sodium concentration of 85 mmol/L
  Interventions: Drug: Furosemide intravenous solution

INTERVENTIONS:
Drug: Furosemide intravenous solution — Diuretics will be titrated to achieve a urine sodium concentration of 50 mmol/L
  Other Names: Lasix
  Arms: 50 mmol/L urine sodium
Drug: Furosemide intravenous solution — Diuretics will be titrated to achieve a urine sodium concentration of 85 mmol/L
  Other Names: Lasix
  Arms: 85 mmol/L urine sodium
Drug: Furosemide intravenous solution — Standard of care
  Other Names: Lasix
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if increasing the dose of diuretics to achieve a higher urine sodium target produces better clinical results when treating patients hospitalized with acute heart failure when compared to lower urine sodium target and standard of care.

The main questions it aims to answer are:

1. Does targeting a higher urine sodium goal achieve greater natriuresis and diuresis?
2. Does targeting a higher urine sodium goal reduce frequency of hospital readmissions?
3. Does targeting a higher urine sodium goal reduce hospital length of stay?

Researchers will compare natriuresis-guided arms with standard of care to see if targeting higher natriuresis goals improves significantly over current practice.

Participants will submit urine samples at routine intervals after being given diuretics to evaluate urine sodium concentration. If urine sodium is low then diuretic dose will be increased.

DETAILED DESCRIPTION:
Patients will be randomized into one of three groups: 50 micromolar natriuresis, 85 micromolar natriuresis, and standard of care. The natriuresis arms will have urine sodium assessed two to four hours administration of intravenous diuretics. If the natriuretic response is inadequate they will immediately receive a higher dose of diuretic. This process will be repeated for the first 72 hours of admission.

ELIGIBILITY:
Inclusion Criteria:

* The study will target adults 18 years of age or older admitted to Lakeland Regional Medical Center who:

  * Have a primary diagnosis of acute decompensated heart failure, and
  * Have at least one of the following signs of hypervolemia:

    * Bilateral lower extremity pitting edema
    * Jugular venous distension
    * Hepatojugular reflex
    * Crackles on pulmonary exam, or
    * Chest x-ray demonstrating pulmonary edema or pleural effusions

Exclusion Criteria:

* Exclusion criteria include:

  * Admission to the intensive care unit
  * Presence of ST-elevated myocardial infarction
  * Presence of type 1 non-ST elevated myocardial infarction
  * Dyspnea primarily due to non-cardiac cause as judged by the emergency medicine physician or admitting physician
  * Use of supplemental oxygen totaling at least 3 L per minute or greater at baseline
  * Anuria
  * End-stage renal disease per KDIGO criteria
  * Dialysis use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Natriuresis at 24 hours | 24 hours
  24-hour natriuresis as measured by urine sodium in a 24-hour urine collection

SECONDARY OUTCOMES:
Natriuresis at 48 hours | 48 hours after enrollment in trial
  Total urine sodium assessed by 24-hour urine collection
Diuresis at 24 hours | 24 hours after enrollment
  Total urine volume assessed by 24 hour collection
Diuresis at 48 hours | 48 hours after enrollment
  Total urine volume assessed via 24-hour collection
Length of Stay | From the date and time of admission order until the date and time of discharge order, assessed for each participant up to 30 days after admission or death from any cause, whichever comes first.
  Duration of hospitalization
Readmission of any cause at 30 days | 30 days after discharge
  Proportion of participants who experience an unplanned hospital readmission for any cause within 30 days after the index hospital discharge.
Readmission rate of any cause at 90 days | 90 days after the time of discharge
  Proportion of participants who experience an unplanned hospital readmission for any cause within 90 days after the index hospital discharge.
Readmission rate of Heart failure | 30 days
  Proportion of participants who experience an unplanned hospital readmission specifically for heart failure within 30 days after the index hospital discharge.
Readmission rate for heart failure | 90 days
  Proportion of participants who experience an unplanned hospital readmission specifically for heart failure within 90 days after the index hospital discharge.
Weight change | Weight assessed at baseline within 24 hours of hospital admission and at discharge, with the discharge weight measured on the discharge day up to 30 days after admission.
  Difference in weight from admission compared to discharge
Net fluid balance | Net fluid balance assessed from baseline Day 1 of admission through hospital discharge, with discharge assessment on the discharge day up to 30 days after admission.
  Cumulative difference between total fluid intake and output during the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lurie, DO, Study Director — Lakeland Regional Hospital; Anas Bizanti, MD, Principal Investigator — Lakeland Regional Hospital
Locations (1):
- Lakeland Regional Hospital, Lakeland, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Yes